CLINICAL TRIAL: NCT04179773
Title: Prospective Observational Study Studying the Influence of the Presence of Liver Cirrhosis During Chemotherapy for ENT Cancer, Upper Digestive Tract Cancer or Colorectal Cancer.
Brief Title: Chemotherapy and Liver Cirrhosis in Frequently-associated Cancers
Acronym: CHIMIOSE
Status: Terminated | Type: Observational
Why Stopped: lack of inclusion
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2018_41; 2018-A01781-54 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Cirrhosis; Neoplasms
Keywords: Liver cirrhosis; chemotherapy; ENT cancers; upper-digestive tract cancers; colorectal cancers
MeSH Terms: conditions — Fibrosis; Neoplasms; Liver Cirrhosis; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cirrhotic patients: Current care study. Data collection on oncological efficacy (Clinical, biological, imaging) Data collection on hepatology (clinical, biological, imaging)
  Interventions: Other: Current care study
- Non-cirrhotic patients: Current care study. Data collection on oncological efficacy (Clinical, biological, imaging) Data collection on hepatology (clinical, biological, imaging)
  Interventions: Other: Current care study

INTERVENTIONS:
Other: Current care study — Observational study in two parts:
  1. Cross-sectional study of patients with digestive or ENT cancer with indication for conventional chemotherapy treatment according to management guidelines, the objective of which is to determine the frequency of cirrhosis.
  2. Exposed/non-exposed cohort study of patients receiving a first course of conventional chemotherapy initiated in outpatient oncology clinic. (safety population).
  Exposed subjects will be patients with cirrhosis, included consecutively. Non-exposed subjects will be non-cirrhotic patients. They will be selected non-consecutively according to the following criteria, for matching to exposed subjects: age (±5 years), type of cancer (digestive vs. ENT), treatment stage (curative vs. palliative). Two unexposed subjects will be selected for 1 exposed subject.

SUMMARY:
Cirrhosis and cancers of the upper digestive tract, colorectal and ENT share common risk factors. Liver cirrhosis can change the elimination of cancer drugs.

Precise data on management and outcome of patients with liver cirrhosis undergoing chemotherapy are lacking. Most patients have been excluded from clinical trials evaluating conventional therapies.

The study of tolerance, side effects, and outcome in patients with cirrhosis could help improve chemotherapy management for better tolerance and efficacy.

The main objective is to estimate the frequency of liver cirrhosis among patients evaluated in CPR for ENT, upper digestive or colorectal cancer.

Secondary objective includes the evaluation ofthe impact of cirrhosis on the management of chemotherapy by comparing cirrhotic patients' outcomes with a control group of matched non-cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up for the following cancers: upper digestive sphere (stomach, esophagus, pancreas, bile ducts), colorectal, ENT
* Theoretical indication of conventional chemotherapy based on 5FU, anthracyclins, platinum salts, gemcitabin, taxans, irinotecan or antiangiogenic drugs, anti-EGFR or anti-HER 2 therapies, according to management guidelines
* Beneficiary of a social security system
* Dated and signed non-opposition consent

Exclusion Criteria:

* Other concomitant primary cancer
* Pregnant women
* Patients under guardianship, curatorship or justice protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected are patients with ENT, upper digestive-tract cancer and colorectal cancer from 2 hospitals: the University Hospital of Lille and the Oscar Lambret Centre.
  The study population consists of patients with a theoretical indication of conventional chemotherapy according to the usual guidelines for the management presented in multidisciplinary board.
  Prospective follow-up will be carried out on the population of patients receiving effective administration of a first course of chemotherapy.
  Patients in theoretical indications who are not receiving chemotherapy will be included in the first part of the study, but prospective follow-up will not be performed in this population.
  Exposed subjects who have received a first course of chemotherapy will be followed prospectively.
  Non-exposed subjects will be matched according to age (+/-5 years), ECOG/WHO classification, chemotherapy protocol and tumour location and followed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with ENT, upper digestive-tract or colorectal cancer with a diagnosis of cirrhosis | before the chemotherapy initiation, within 45 days of multidisciplinary board

SECONDARY OUTCOMES:
Percentage of patients receiving at least a first effective course of chemotherapy on all patients with a theoretical indication for chemotherapy | within 45 days of multidisciplinary board.
Survival time | the date of death, the date of last news or the point date (12 months).
  Survival time defined as the difference between the date of initiation of chemotherapy,
Progression-free survival time | the date of initiation of chemotherapy, tthe date of progression or death, the date of last news or the point date (12 months).
  Progression-free survival time defined as the difference between the date of initiation of chemotherapy, the date of progression or death, the date of last news or the point date (12 months).
Frequency of chemotherapy side effects according to CTCAE version 5.0 classification in cirrhotic patients who have received chemotherapy | Up to 5 years after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Massih Ningarhari, MD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille
  - Hôpital Claude Huriez, CHU, Lille